CLINICAL TRIAL: NCT07104279
Title: Multicenter, Post-Market Clinical Follow-up Study of the Z1 Femoral Hip System
Brief Title: Z1 Hip System: Post-Market Clinical Follow Up Study
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2024-25H
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hip Osteoarthritis; Acute Traumatic Fracture of the Femoral Head or Neck; Avascular Necrosis of the Femoral Head
Keywords: total hip arthroplasty; total hip replacement; osteoarthritis; hemiarthroplasty; partial hip replacement
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects implanted with the Z1 Femoral Hip System
  Interventions: Device: Z1 Femoral Hip System

INTERVENTIONS:
Device: Z1 Femoral Hip System — Subjects who will be implanted with the Z1 Femoral Hip System in hemi-hip arthroplasty and primary total hip arthroplasty

SUMMARY:
The objectives of this study are to confirm the early to mid-term safety, performance, and clinical benefits of the Z1 Femoral Hip System in hemi-hip arthroplasty and primary total hip arthroplasty.

The primary objective of this post market clinical follow-up (PMCF) study is the assessment of safety by recording and analyzing the survival of the implant system at 2 years post-implantation. Safety will also be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to implant, instrumentation, and/or procedure should be specified.

The secondary objective is the assessment of functional performance and clinical benefits of the Z1 Femoral Hip System demonstrated by recording patient-reported clinical outcomes measures (PROMs).

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a common operative treatment where an arthritic, degenerative or fractured hip joint is replaced with a prosthetic device if conservative options are unable to relief pain and debilitating symptoms. A femoral stem component is used in conjunction with a femoral head component for the replacement of the proximal femur in total hip or hemi hip arthroplasty. THA now includes young and active patients, as well as very old ones thanks to the continuous improvement in implant design. Major indications include osteoarthritis, rheumatoid arthritis, avascular necrosis (AVN) and hip fractures. The surgical procedure consists in replacing the head of the femur and acetabulum (socket) with a prosthesis. Another type of hip arthroplasty is called Hemi arthroplasty, which does not include the replacement of the acetabulum.

This system is composed of a femoral stem that is inserted into the femoral canal, a ball that attaches to the femoral stem, and an acetabular component or shell that replaces the acetabulum. Device components are made from durable materials that can withstand loads applied to the artificial hip joint during physical activity, are resistant to corrosion and fatigue, provide minimal friction and wear, and are biocompatible. Commonly used materials include cobalt chrome, commercially pure titanium, titanium alloy with aluminum and vanadium, ceramics, and ultrahigh molecular weight polyethylene.

Clinical studies have proven implant longevity in both cementless and cemented THA, offering patients effective long-term relief. In cementless THA, successful biological fixation is dependent on bony on-growth onto the surface of the prosthesis whereas, cemented fixation depends on a stable interface between prosthesis and cement and a solid mechanical bond between cement and bone. Ultimately, the goal of a THA is to bring the patients back to their normal routine without pain and stiffness. THA and hemiarthroplasty are both very successful procedures with an 84-97% patient satisfaction rate and an implant survival of over 90% after 10 years (THA) and implant survival of approximately 93% at 10 years (Hemiarthroplasty).

The Z1 Femoral Hip System consists of femoral hip stems intended for use in total or hemi hip arthroplasty. The triple-tapered stem is designed for implantation into the proximal femur and mates with compatible femoral heads and adapters for use in total or hemi hip arthroplasty through a 12/14 male taper connection.

The stems are manufactured from a forged titanium alloy Ti-6Al-4V and have a wedge-shaped design, with a proximal-to-distal taper. Apart from the highly polished femoral neck region, the entire surface of the stem is gritblasted and sprayed with a Ti-6Al-4V titanium alloy plasma coating followed by a hydroxyapatite (HA) overcoat. Offered in multiple sizes and neck lengths, the stems are available in Standard, High Offset, and Coxa Vara offsets to accommodate various patient anatomies. The hip stems are provided sterile and are for single use only. System-specific instrumentation is available to prepare the femur for implantation of the Z1 Hip System femoral stems. The Z1 Hip System is for use only with the Zimmer Biomet femoral heads and adapters, bipolar heads, and acetabular shells and liners identified in the package insert as compatible components.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old and skeletally mature
* Patient is physically and mentally willing and able, in the Investigator's opinion at the time of enrollment, to be compliant with the protocol, including all scheduled study evaluations
* Patient, or the patient's legally authorized representative, is willing and able to participate in the Informed Consent process and provide their consent
* Independent of study participation, patient is a candidate and qualifies for primary total hip or hemi-arthroplasty based on physical exam and medical history including at least one of the following:

  * Advanced wear of the joint due to degenerative, post-traumatic or rheumatic diseases
  * Acute traumatic fracture of the femoral head or neck
  * Avascular necrosis (AVN) of the femoral head

Exclusion Criteria:

* Revision arthroplasty
* Acute, chronic, local, or systemic infection(s)
* Severe muscular, neural, or vascular diseases that endanger the limb(s) involved
* Lack of bony structures proximal or distal to the joint, so that good anchorage of the implant is unlikely or impossible
* Total or partial absence of the muscular or ligamentous apparatus
* Any concomitant diseases that can jeopardize the functioning and the success of the implant
* Allergy to the implanted material, especially to metal (e.g. cobalt, chromium, nickel, etc.)
* Local bone tumors and/or cysts
* Patient has any condition that would, in the Investigator's opinion, place the patient at undue risk or interfere with the study
* Any vulnerable subject:

  * a prisoner
  * a patient known to be pregnant
  * mentally incompetent or unable to understand what participation in the study entails
  * a known substance abuser

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should consist of up to 150 subjects implanted with the Z1 Femoral Hip System in hemi or total hip arthroplasty, according to the approved indications.
  Inclusion and exclusion criteria are based on the indications and contraindications defined in the IFU for the Z1 Femoral Hip System.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
2 Year Survivorship | 2 years post-operative
  The absence of removal of the study device will be evaluated using Kaplan Meier method. The safety of the system will additionally be assessed by monitoring the frequency and incidence of adverse events, including relation to implant, instrumentation, and/or procedure.

SECONDARY OUTCOMES:
HOOS JR | 5 years post-operative
  The functional performance and clinical benefits of the study device will be assessed by a patient-reported clinical outcomes measure (PROM)(HOOS JR).

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - OrthoCarolina/OrthoCarolina Research Institute, Charlotte, North Carolina
  - Orthopedic & Fracture Specialists, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided